CLINICAL TRIAL: NCT04749628
Title: Effects of Cannabidiol (CBD) Oral Solution in Patients Undergoing Bilateral Total Knee Arthroplasty: a Randomized, Controlled, Parallel, Triple Blind, Pilot Study
Brief Title: Cannabidiol for Bilateral Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-1688
Record Dates: First submitted 2021-02-05; First posted 2021-02-11 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-10

CONDITIONS: Pain, Postoperative; Opioid Use; Knee Osteoarthritis
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Knee | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ora-sweet SF (Placebo Comparator)
  Interventions: Other: Ora-sweet SF
- 400mg cannabidiol (Experimental)
  Interventions: Drug: cannabidiol
- 800mg cannabidiol (Experimental)
  Interventions: Drug: cannabidiol

INTERVENTIONS:
Drug: cannabidiol — Epidiolex (cannabidiol) oral solution
  Other Names: Epidiolex
  Arms: 400mg cannabidiol; 800mg cannabidiol
Other: Ora-sweet SF — Ora-sweet SF placebo
  Arms: Ora-sweet SF

SUMMARY:
In light of the opioid epidemic and evidence suggesting that cannabis may be opioid-sparing, we are in a unique position to conduct a novel, high-impact study that would set the stage for future RCTs examining the effects of a nonintoxicating and nonaddictive cannabinoid in an orthopedic patient population. Epidiolex®, an oral cannabidiol (CBD) solution, is the first ever cannabis-derived medication to be approved by the Food & Drug Administration. Our aim is to conduct a pilot study using a placebo oral solution, 400mg and 800mg Epidiolex® to gather data on its effects on patients undergoing bilateral total knee arthroplasty (BTKA). We will be estimating whether Epidiolex® is associated with minimal opioid use and adequate analgesia. We will also assess its tolerability, pharmacokinetics, and effects on inflammatory markers in the perioperative setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75
* Scheduled for same-day bilateral total knee replacements with participating surgeons
* American Society of Anesthesiologists (ASA) Physical Status 1 or 2

Exclusion Criteria:

* ASA 3 and higher
* Weight < 40kg
* Planned use of general anesthesia
* Contraindication to major components of study protocol
* Cannabis or cannabinoid use within the past 3 months (recreational and/or medical)
* Use or ingestion of hemp seeds or hemp oil in any form within the past 30 days
* Chronic opioid use (>3 months)
* Coumadin use
* Current use of SSRI or SNRIs
* History of substance abuse or dependence
* Active or history of major psychiatric illness
* Severe cardiovascular disorder
* Severe hepatic or renal insufficiency (transaminase levels above ULN)
* History of epilepsy
* Diagnosis of rheumatic disease, autoimmune disease, or immunodeficiency (e.g. rheumatoid arthritis, psoriatic arthritis, inflammatory bowel disease, multiple sclerosis, etc.)
* Use of valproate or clobazam
* Known or suspected hypersensitivity, allergy, or contraindication to cannabinoids or any of the excipients in the study medications (i.e. sesame oil, sucralose, strawberry flavor)
* Active use of steroids - oral steroids upon admission
* Stress dose steroids
* Non-English speakers
* Planned discharge to home without caregiver(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Cumulative Opioid Usage in First 72 hours Postoperatively | 0-72 hours postoperatively
  Cumulative opioid usage over the first 72 hours after surgery. Measured in morphine equivalents (ME), a scale that measure opioid usage among all opioid medications

SECONDARY OUTCOMES:
Pharmacokinetics of CBD | 0, 1, 2, 3, 4, 6 hours after medication administration
  Levels of CBD in the blood. This is measured using blood draws and lab analysis.
Levels of Plasma Inflammatory Marker Interleukin-6 | Preoperative, Postoperative day 1
  Interleukin-6 (IL6) is an inflammatory marker found in plasma. The levels of IL6 are measured using blood draws and lab analysis.
NRS Pain at rest | Preoperatively; postoperatively in the PACU, morning of postoperative day (POD) 1,2,3,4,7 and at 3 months
  Pain at rest measured using numerical rating scale(NRS) from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
NRS Pain with movement | Preoperatively; morning of postoperative day (POD) 1,2,3,4,7 and at 3 months
  Pain with movement using numerical rating scale(NRS) from 0-10, with 0 being no pain at all to 10 being the worst pain imaginable.
Brief Pain Inventory Short Form | Preoperatively; morning of postoperative day (POD) 1,2,3,4,7 and at 3 months
  Brief Pain inventory short form measures the severity of pain and its impact on function. It measures pain from 0-10 0 being no pain whatsoever to 10 being the worst pain imaginable. It measures impact on function from 0-10, 0 being no impact whatsoever to 10 being completely impactful.
Incidence of adverse events | Postoperatively in the PACU; morning of postoperative day (POD) 1,2,3,4,7 and at 3 months
  Adverse events, including allergic reactions, pyrexia (fever), somnolence (excessive sleepiness), GI problems (upset stomach, diarrhea), dry mouth, escalation of post-operative opioid requirement
Opioid related Symptom Distress Scale (ORSDS) | Morning of postoperative day (POD) 1,2,3,4,7 and at 3 months
  ORSDS measures opioid related side effects. There are 13 side effects with 3 subcategories (severity, frequency, bothersomeness) each with 5 different responses (scored 0-4).
Anxiety levels | Preoperatively; Morning of postoperative day (POD) 1,2,3,4,7 and at 3 months
  Hospital Anxiety and Depression Scale (HADS) asks 14 questions, 7 about anxiety and 7 about depression. Responses are scored from 0-3. Responses between the two categories are summed and scoring is as follows: 0-7 = normal, 8-10=borderlines abnormal, 11-21=abnormal
Cumulative inpatient analgesic use (non-opioid) | POD0 - POD3
  Total non-opioid medication usage
Opioid & non-opioid analgesic consumption | At hospital discharge to POD7 and at 3 months
  Total opioid & non-opioid medication usage
Hospital length of stay | End of surgery to hospital discharge
  Length of stay measured in hours
Blinding Assessment | POD4
  Patients are asked which treatment they think they received. The correctness of their guesses is then measured using the bang-blinding index to see if patients were able to accurately guess which treatment they received. It is measured on a scale of -1 to 1. Scores closer to 0 indicate better blinding, or patients not being able to guess their treatment
Time to reach discharge physical therapy goals | At hospital discharge - up to 3 days after surgery
  Physical therapy goals for total knee replacement include walking 100 feet, going up and down 4 stairs, and independent transfer (meaning they can move from a lying to standing position independently). Patients need to complete these goals before being discharged
Range of motion | preoperatively, 6 weeks postoperatively.
  Range of motion, or extension and flexion of the knees, are measured preoperatively and at the patients' 6 week surgeon visit. It is measured in degrees
Sleep quality and duration | POD0 - POD3
  Sleep quality assessed by actigraphy using ActiGraph wGT3X-BT activity monitor
Sleep quality | preoperatively; morning of postoperative day (POD) 1,2,3,4,7 and at 3 months
  Sleep quality assessed by Leeds sleep evaluation questionnaire (LSEQ). Responses to 10 questions will be measured on a slider scale ranging from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Sideris, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: For researchers who provide a methodologically sound proposal and analyses to achieve aims in the approved proposal. Proposals should be directed to siderisa@hss.edu. To gain access, data requestors will need to sign a data access agreement.